CLINICAL TRIAL: NCT00969839
Title: A Study to Evaluate the Safety and Effectiveness of the NovaLign Intramedullary Fixation System for the Treatment of Humeral Diaphysis Fractures
Brief Title: NovaLign Intramedullary Fixation System (IFS) for the Treatment of Humeral Fractures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NovaLign Orthopaedics, Inc (Industry)
Responsible Party: Dawn Norman, Director, Clinical Affairs, NovaLign Orthopaedics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-001
Record Dates: First submitted 2009-08-30; First posted 2009-09-01 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Fracture
Keywords: Fracture; Humerus; Intramedullary; Fixation
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intramedullary Fixation System (Experimental): Humeral fractures to be treated with the Intramedullary Fixation System
  Interventions: Device: NovaLign Intramedullary Fixation System

INTERVENTIONS:
Device: NovaLign Intramedullary Fixation System — Intramedullary fixation of broken humerus

SUMMARY:
This post-market clinical study is being done to evaluate the use of the NovaLign™ Intramedullary Fixation System in the treatment of humeral fractures.

DETAILED DESCRIPTION:
This is an observational, prospective, nonrandomized open label, post-market clinical study, designed to evaluate the use a flexible intramedullary fixation device used in the treatment of fractures of the humerus. This is a multicentre trial.

ELIGIBILITY:
Inclusion Criteria:

* Humeral Fracture
* Surgical intervention can be performed within 14 days of injury (injury being Day 0 for this particular criteria)
* Fully functioning contralateral limb (e.g., hand, arm, shoulder)
* Age 18 years or older and skeletally mature

Exclusion Criteria:

* Intraarticular fractures or those involving shoulder or elbow of the index arm
* Pathologic fracture (e.g., tumor involvement, osteomalacia, etc.; osteoporosis is not an exclusion)
* Evidence of neurologic injury in the index arm, including compartment syndrome or radial nerve palsy
* Additional upper body injuries (e.g., upper extremity, abdominal, thoracic, neck or head injury) that may affect or inhibit the evaluation of the index or contralateral arm, shoulder, elbow, etc or would not allow the patient to follow or comply with appropriate post-operative regimens
* Any previous bodily injury or surgery that may interfere with function or evaluation of index or contralateral arm, shoulder, elbow, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Radiographic union and safety | 12 months

SECONDARY OUTCOMES:
Function, pain, and quality of life assessments at regular intervals | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: B Crist, MD, Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - Denver Health Medical Center, Denver, Colorado
  - University of Missouri - Columbia, Columbia, Missouri